CLINICAL TRIAL: NCT06199674
Title: Effects of Photobiomodulation Therapy (PBM) on Dental and Periodontal Health of Patients Undergoing Fixed-appliance Orthodontic Treatment
Brief Title: Effects of PBM on Fixed-appliance Orthodontic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zhiyi Shan, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PBMRR-HKU-143
Record Dates: First submitted 2023-12-01; First posted 2024-01-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Orthodontics; Root Resorption
Keywords: photobiomodulation; fixed-appliance orthodontic treatment; root resorption; orthodontic pain; tooth movement
MeSH Terms: conditions — Root Resorption | interventions — Low-Level Light Therapy; Orthodontic Appliances, Fixed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PBM group (Experimental): wear PBM device daily during the fixed-appliance orthodontic treatment
  Interventions: Device: photobiomodulation therapy; Other: orthodontic fixed-appliance
- Control group (Sham Comparator): wear sham device daily during the fixed-appliance orthodontic treatment
  Interventions: Other: orthodontic fixed-appliance

INTERVENTIONS:
Device: photobiomodulation therapy — Patients in the PBM group will be delivered a portable PBM device (PBM Healing Ortho) at the beginning of orthodontic treatment and will be instructed to use it daily at home for 8 minutes (4 min per arch) after tooth brushing.
  Arms: PBM group
Other: orthodontic fixed-appliance — All eligible patients will receive orthodontic treatment with a pre-adjusted fixed appliance (0.022'' × 0.028'' slot system, MBT, 3M Unitek) provided by the same practitioner. At the start of treatment, a cantilever auxiliary arch bent with a 0.017'' × 0.025'' Stainless Steel wire (3M Unitek) will be used to apply a 100 g intrusion force to the premolars that will be extracted in 3 months. All other teeth will undergo regular orthodontic treatment with a standard archwire protocol (0.014'' NiTi, 0.016'' NiTi, 0.018'' NiTi, 0.017'' × 0.025'' NiTi, 0.019'' × 0.025'' NiTi, and 0.019'' × 0.025'' SS, 0.019'' × 0.025'' TMA) for alignment, leveling, space closure, detailing, and finishing. For en masse retraction, a 150 g force will be applied by coil springs, allowing bracket slots to slide along the 0.019'' × 0.025'' SS.

SUMMARY:
The aim of this study is to investigate the effects of photobiomodulation therapy (PBM) on the dental and periodontal health of patients undergoing fixed-appliance orthodontic treatment, including orthodontically induced root resorption, orthodontic pain, space closing rate, and dental microbiome profile in dental plaques.

DETAILED DESCRIPTION:
Photobiomodulation therapy (PBM) is a non-invasive, adjunctive medical treatment that has promising effects on various dental and oral conditions, including controlling inflammation, promoting wound healing, and relieving pain. While animal studies have explored PBM therapy in orthodontics for accelerating tooth movement, preventing root resorption, alleviating pain, and controlling periodontal inflammation, clinical studies with high-quality evidence remain limited. Therefore, a randomized controlled trial (RCT) will be conducted to investigate the effects of a portable PBM device on the dental and periodontal health of patients undergoing fixed-appliance orthodontic treatment. This two-arm RCT will be conducted with a triple-blinded and parallel study design in a 1:1 ratio. Fifty orthodontic patients will be recruited at the Prince Philip Dental Hospital following the eligibility criteria from Jan. 2024 to Jan. 2026 (24 months) and evenly distributed to the two arms. Randomization and allocation will be conducted by a statistician who will not participate in the intervention and outcome assessment process using computer software. Participants in the PBM group will be required to wear a PBM device, while those in the control group will receive a sham device with an identical appearance to the PBM device but without light irradiation. All participants must wear their assigned device daily for 8 minutes (4 minutes for the upper and lower dental arches each) after brushing their teeth during the process of fixed-appliance orthodontic treatment. The allocation sequences will be concealed in a batch of opaque envelopes. Patients and the outcome assessor will be blinded to the allocation sequence. This protocol is proposed in compliance with the Declaration of Helsinki and the ICH-Good Clinical Practice (GCP) Guideline. The study will be conducted and reported according to the Consolidated Standards of Reporting Trials (CONSORT) guideline. Written consent will be obtained from all subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 and 35 years old with permanent dentition
2. Patients who undertake orthodontic treatment using fixed appliances
3. Patients who require extraction of premolars in either their upper or lower dental arch
4. Patients who have fair oral hygiene habits
5. Patients who are systemically healthy

Exclusion Criteria:

1. Patients with generalized dental caries and severe chronic periodontitis in stages III and IV
2. Patients with congenital or severe craniofacial anomalies which necessitate orthognathic surgery
3. Patients with physical or mental impairment, and those who smoke or undertake systemic medications
4. Patients with current root resorption at any of the teeth
5. Patients with endodontic treatment and/or large restorations on premolars to be extracted

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Orthodontic-induced inflammatory root resorption (OIIRR) | baseline, 3 months after intrusive force loading
  Record OIIRR by calculating the volume of craters on the root surfaces of the extracted tooth using a standard micro-CT machine after 3 months following intrusions by cantilever auxiliary arch.

SECONDARY OUTCOMES:
Orthodontic pain | baseline, immediately after fixed appliance placement and immediately after adjustment every month during the first year of regular orthodontic treatment
  Record orthodontic pain monthly since the beginning of regular orthodontic treatment by patients' self-registration on a 100-millimetre Visual Analogue Scale (VAS). 0 means "no pain", 100 means "worst pain", the higher the score, the more severe the pain. In addition, 5-millilitre unstimulated saliva samples will be collected from each participant with the same time scheme for evaluation of pain-related biomarkers.
Space closure by en masse retraction | every month from the start of space closure to the end of closure, taking into account the very slow closure of space, assessed up to 12 months
  Record the duration of the space closure by calculating the rate of tooth movement (mm/mo) with physically measurement. In addition, gingival crevicular fluid samples will be collected from the two space-neighbouring teeth to analyse bone-related biomarkers.
Microbiome profile in dental plaques | baseline, every 3 months from the start of regular orthodontic treatment to the end of treatment process
  Samples of supragingival and subgingival plaques will proceed to 16S rRNA sequencing for analysis of microbiome profiles, and q-PCR for evaluating bacterial loads of some critical pathogens for dental caries and periodontitis.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyi Shan, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong